CLINICAL TRIAL: NCT00768950
Title: The Characterization of Small Bowel and Colonic Involvement in Patients With Seronegative Spondyloarthritides
Acronym: SPONDILENDO
Status: Completed | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Collaborators: EXECUTIVE UNIT FOR FINANCING HIGHER EDUCATION AND SCIENTIFIC UNIVERSITY RESEARCH (Unknown); Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, Prof. Dr. Mihail Radu Voiosu, University Professor, Carol Davila University of Medicine and Pharmacy
Other Study IDs: UMFCD-Idei-320/2007; Idei-320/01-10-2007
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Spondyloarthropathies
Keywords: Seronegative spondyloarthropathies; Endoscopic capsule examination; Small bowel and colon lesions; Nonsteroidal anti-inflammatory drugs; Anti TNF Alpha Drugs
MeSH Terms: conditions — Spondylarthropathies | interventions — Infliximab; Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Spondyloarthropathies: Patients with spondyloarthropathies (ankylosing spondylitis, reactive arthritis, psoriatic arthritis and spondylitis, enteropathic arthritis and spondylitis, juvenile-onset spondyloarthritis, and undifferentiated spondyloarthritis) as defined by the AMOR criteria
  Interventions: Procedure: Capsule endoscopy examination; Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Capsule endoscopy examination — Examination of the small bowel with endoscopic videocapsule
  Other Names: Given imaging capsule SB2
Procedure: Colonoscopy — Endoscopic examination of the large bowel and terminal ileum
  Other Names: Olympus Evis Exera II videocolonoscope

SUMMARY:
Up to 60% of patients with Seronegative Spondyloarthritides have inflammation in the colon or ileum. This is usually asymptomatic, but in 5 to 10% of patients with SA, Frank IBD will develop. Lesions of the bowel could also be present in the SA patients because of the potential injury posed by the NSAIDS, a common used medication in this setting.

It is the bowel involvement in patients with SA that we propose to characterize, partly because there are scant communicated data in the medical literature, especially regarding small bowel lesions.

DETAILED DESCRIPTION:
The Seronegative Spondyloarthritides (SA) are a group of disorders that share certain clinical features and an association with the hla-b27 allele, having also overlapping features with inflammatory bowel disease (IBD).

Up to 60% of patients have inflammation in the colon or ileum. This is usually asymptomatic, but in 5 to 10% of patients with SA, Frank IBD will develop.

Lesions of the bowel could also be present in the SA patients because of the potential injury posed by the NSAIDS, a common used medication in this setting.

On the other hand, biologics used to treat patients with SA are believed to favorably influence the small bowel lesions that are concomitantly present.

It is the bowel involvement in patients with SA that we propose to characterize, partly because there are scant communicated data in the medical literature.

The design of the proposed study involves performing one full colonoscopic examination (including ileoscopy) followed by one capsule endoscopy examination to the patients with SA. Prior to these examination, the patency of the gi tract will be tested using a patency capsule. If the patency of the gi tract is not confirmed, then the capsule endoscopy examination is abandoned.

Our aim is to explore about 100 patients in three years, thus having a close-to-reality "look" into the presence and extent of bowel involvement in the pool of the patients having SA; and also to characterize the lesions mainly depending on the treatment received, concomitant pathology and the form of the disease. We also aim to identify a relationship between the lesions found at colonoscopy and capsule endoscopy, the purpose being the possibility to predict one having only performed the other.

Thus, we hope to identify the therapeutic strategies that are most suited in the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* signing of the inform consent
* subjects 18 years old or more
* patients with spondyloarthropathy as defined by the Amor criteria

Exclusion Criteria:

* presumed intestinal obstruction
* impaired deglutition
* cardiac pace-makers present
* pregnancy
* pelvic or abdominal radiotherapy anytime in the past
* major abdominal surgery anytime in the past
* major comorbidities which could represent a contraindication to a surgical abdominal intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spondyloarthropathies (ankylosing spondylitis, reactive arthritis, psoriatic arthritis and spondylitis, enteropathic arthritis and spondylitis, juvenile-onset spondyloarthritis, and undifferentiated spondyloarthritis) reffered to a Universitary Clinic of Internal Medicine and Rheumatology
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2008-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with bowel lesions | July 2012

SECONDARY OUTCOMES:
Correlation of the bowel lesions with patient status | July 2012

CONTACTS AND LOCATIONS:
Overall Officials: Mihail R Voiosu, M.D., Ph.D., Principal Investigator — Carol Davila University of Medicine and Pharmacy; Mihai Rimbas, M.D., Study Chair — Carol Davila University of Medicine and Pharmacy
Locations (1):
- Gastroenterology Department, Colentina Clinical Hospital, Bucharest, Romania

REFERENCES:
- [Background] Rimbas M, Marinescu M, Voiosu MR. Bowel lesions in spondyloarthritides. Rom J Intern Med. 2009;47(1):75-85. PMID 19886073
- [Result] Rimbas M, Marinescu M, Voiosu MR, Baicus CR, Caraiola S, Nicolau A, Nitescu D, Badea GC, Parvu MI. NSAID-induced deleterious effects on the proximal and mid small bowel in seronegative spondyloarthropathy patients. World J Gastroenterol. 2011 Feb 28;17(8):1030-5. doi: 10.3748/wjg.v17.i8.1030. PMID 21448355
- [Derived] Chitul A, Voiosu AM, Marinescu M, Caraiola S, Nicolau A, Badea GC, Parvu MI, Ionescu RA, Mateescu BR, Voiosu MR, Baicus CR, Rimbas M. Different effects of anti-TNF-alpha biologic drugs on the small bowel macroscopic inflammation in patients with ankylosing spondylitis. Rom J Intern Med. 2017 Mar 1;55(1):44-52. doi: 10.1515/rjim-2017-0001. PMID 28103201